CLINICAL TRIAL: NCT01117493
Title: Expert Patient Self-management Programme Versus Usual Care in Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Dr Judy Bradley, Belfast Health and Social Care TRust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06054JB-A
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-04

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Other): Usual care included reviews at a specialist respiratory clinic on a three monthly basis to monitor spirometry, inflammatory blood markers and sputum microbiology. The patients were prescribed inhaled therapy and antibiotics if required, and treatment adjusted to the needs of the patient as necessary, including hospital admission.
  Interventions: Behavioral: Usual care
- Expert Patient Programme (Experimental): Receives a disease specific Expert Patient Programme in addition to usual care. The disease specific Expert Patient Programme was delivered one session per week (lasting 2½ hours) for eight weeks and included 2 weeks disease specific education followed by 6 weeks standardised Expert Patient Programme.
  Interventions: Behavioral: Expert Patient Programme

INTERVENTIONS:
Behavioral: Expert Patient Programme — Intervention was a disease specific Expert Patient Programme in addition to usual care. The disease specific Expert Patient Programme was delivered one session per week (lasting 2½ hours) for eight weeks and included 2 weeks disease specific education followed by 6 weeks standardised Expert Patient Programme.
  Other Names: Self-management
  Arms: Expert Patient Programme
Behavioral: Usual care — Usual care included reviews at a specialist respiratory clinic on a three monthly basis to monitor spirometry, inflammatory blood markers and sputum microbiology. The patients were prescribed inhaled therapy and antibiotics if required, and treatment adjusted to the needs of the patient as necessary, including hospital admission.
  Other Names: Usual management
  Arms: Usual care

SUMMARY:
The aim of this exploratory randomized controlled trial was to investigate the efficacy of a disease specific Expert Patient Programme compared to usual care in patients with bronchiectasis. Hypothesis: Disease specific EPP will increase self efficacy compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) with a primary diagnosis of bronchiectasis based on a respiratory physician's assessment including a computed tomography scan were included in the study

Exclusion Criteria:

* Primary diagnosis of cystic fibrosis
* Patients with methicillin-resistant Staphylococcus aureus infection
* Patients with any condition that would have an impact on the assessment procedures (e.g. sensory impairment, pregnancy, language barriers)
* Any factor that would prevent adherence to the self-management programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 8 months
  Self efficacy is measured using the Chronic Disease Self Efficacy Scale. Confidence is measured on a 1-10 point Likert scale for 10 subscales. There are no specific units for this measurement.

SECONDARY OUTCOMES:
Perception of illness | 8 months
  Perception of illness is measured using the Illness Perception Questionnaire - revised IPQ-R. This questionnaire has 8 domains. Minimum score 52 and maximum 204. There are no specific units for this measurement.
Health related quality of life | 8 months
  Health related quality of life is measured using the St Georges Respiratory Questionnaire. This questionnaire has 3 domains. Min-max scores 0-100%
Self rated health | 8 months
  An expert patient programme questionnaire is used to record self rated health, management of condition, days lost to work and social activities, satisfaction and benefits. There are no specific units for this measurement.
Lung function | 8 months
  Spirometric measurement of FEV1 expressed as a percentage predicted is used to assess lung function
Rate of exacerbation | 8 months
  Frequency of antibiotics is recorded to assess rate of exacerbation. These will be expressed as the number of antibiotics prescribed per group during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Judy M Bradley, PhD, Principal Investigator — Belfast Health and Social Care Trust & University of Ulster